CLINICAL TRIAL: NCT07376031
Title: Effect of Thermal Ablation on Persistent HPV Infection in Danish Women ≥40 Years of Age; a Randomized Clinical Study
Brief Title: Cervical Thermal Ablation to Treat Persistent HPV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Jesper Bonde, Senior Researcher, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJ:845; A2971 (Other Grant/Funding Number: Fonden for Faglig Udvikling i Speciallægepraksis)
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cervical Cancer Screening; HPV; Thermal Ablation
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No treatment (No Intervention): Women eligible not receiving thermal ablation
- intervention (Active Comparator): thermal ablation was performed using the WISAP Probe 6004/6005/6002 at 65 degrees Celsius for 2 minutes, and at 100 degrees Celsius for 40 seconds as defined in Danish guidelines. In the absence of visible lesions, the entire transformation zone was treated. For transformation zones extending into the endocervical canal (type 3), treatment was applied to the visible ectocervix, recognizing the technical limitations of thermal ablation for endocervical disease. Ablation treatment was administered as two consecutive treatments 2-3 days apart at the gynecologist´s discretion.
  Interventions: Procedure: Treatment

INTERVENTIONS:
Procedure: Treatment — Thermal ablation was performed using the WISAP Probe 6004/6005/6002 at 65 degrees Celsius for 2 minutes, and at 100 degrees Celsius for 40 seconds as defined in Danish guidelines.
  In the absence of visible lesions, the entire transformation zone was treated. For transformation zones extending into the endocervical canal (type 3), treatment was applied to the visible ectocervix, recognizing the technical limitations of thermal ablation for endocervical disease. Ablation treatment was administered as two consecutive treatments 2-3 days apart at the gynecologist´s discretion.
  Arms: intervention

SUMMARY:
Thermal ablation of women ≥40 years of age with persistent Human papillomavirus (HPV) infection. A pilot and intervention study.

Cervical heat treatment is a relatively new form of treatment19 where a smaller, defined area of the cervix is destroyed by insertion of a heated probe. Cervical heat treatment is already used in specialist medical practice for patients with erythroplakia, contact bleeding, chronic cervicitis and discharged. In a collaboration between Region Zealand and the Capital Region of Denmark, 120 women are randomized to receive thermal ablation for HPV infections without severe disease with a matched control group of 120 women who do not receive ablation. All women are monitored through repeated cervical cytology re-tests at defined follow-up (FU) times. The study cohort consist of 1) sample on enrollment date, 2) 3 months FU sample, 3) 6 months FU sample, 4) 12 months FU sample. All samples are collected in SurePath liquid-based cytology medium and HPV tested using the BD Onclarity HPV test (BD Integrated Diagnostic systems, Sparks, MD)20-22 supplemented by a full genotyping analysis (Seegene, Seoul, Korea)21,23. Methylation status is examined using the QiaSure FAM19A4/miRNA 122-4 methylation test (Qiagen, Hilden, Germany).

This project element aims to determine whether thermal ablation impact viral clearance compared to the control group, and whether DNA methylation status is significant amongst women who are persistently HPV positive before and after thermal ablation.

DETAILED DESCRIPTION:
Persistent infection with high-risk human papillomavirus (HR-HPV) is the etiological cause of precancerous cervical intraepithelial neoplasia (CIN) and ultimately cervical cancer (CC)1. With 50 years of cervical cancer screening in Denmark, CC incidence has been reduced from the peak of 39.6/100.000 in 1966 to 11/100.000 in 20222, but the World Health Organization world elimination goal of 6/100.0003,4 is still in the distance.

Cervical cancer is largely preventable through local treatment of screen-detected cervical precursor lesions also known as cervical intraepithelial neoplasia (CIN). Infection with the HPV virus causes cell changes and cervical cancer5. The HPV virus infects the cells on the surface of the cervix. While most women naturally clear an HPV infection over time, in approx. 10% of all infected women, the HPV infection becomes persistent which is a known risk enhancer6-8. It is unknown why an HPV infection becomes chronic in some but not most women. Lifetime risk of HPV infection is over 80%. In Denmark, all women between 23-65 years are offered screening for cervical cancer at defined intervals. Today, cervical screening is conducted using a combination of cell-based evaluation, cytology, and molecular HPV screening. However, Danish cervical cancer screening is in transit from cytology to molecular HPV based screening to all women aged 30 to 649. A recurrent issue with HPV based screening is the specificity of the screening which leads to many women being referred for monitoring or follow up without having significant disease. The screening program constitute 400,000 individual annual screening samples and approx. 30,000 tissue biopsy sets are derived as follow-up after a positive screening sample. From these, 6500 cone sections results.

Cervical cancer incidence in Denmark displays a double peaked pattern with the highest incidence in women 35-45 years and again in women 70-75 years. The latter peak is closely related to the current exit age from screening which is 64 years compared to 70 in the other Nordic countries. From 2012-2016, the average annual number of new CCs was 371 with 103 annual deaths10. In Denmark, women aged ≥ 60 years accounts for more than half of CC deaths (66%) and almost 30% of new cases10. For older women as well as younger, a clinical challenge is that many carry a persistent HPV infection which may or may not give rise to severe dysplasia possibly preceding cancer. However, current diagnostic methodologies offer no safe way to distinguish between the progressive lesions and persistent, non-progressive HPV infections. This leads to a large group of persistent HPV positive women in extended clinical follow-up regimens without a clear exit strategy and eventually leading to (over)treatment in the form of conization or hysterectomy. DNA methylation of human genes has shown to be particularly sensitive for the detection of cervical cancer and advanced CIN2 or 3 and presumed increased short-term risk of progression to cervical cancer11-17. Absence of host-cell DNA methylation on the other hand, is associated with regression of CIN2/313,17.

This PhD project focusses on whether novel methylation biomarkers can assist in risk-stratification for risk of severe cervical disease in two groups of women with persistent human papillomavirus (HPV) infections:

* Women who have received thermal ablation as part of treatment for non-severe cell changes following HPV infection (randomized control trial, Region Zealand)
* Women 60-64 years of age with persistent HPV infections participating in cervical cancer screening in the Capital Region of Denmark If successful, the project will provide needed data to support introduction of molecular triage biomarkers in two different applications; to determine persistent HPV infection after thermal ablation treatment and to risk stratify women aged 60-64 years before conclusion of screening program participation18. The project is a collaboration between 1) Region Zealand and Capital Region of Denmark, and 2) Capital Region of Denmark and Central Denmark Region.

Project element 1: Thermal ablation of women ≥40 years of age with persistent HPV infection. A pilot and intervention study.

Cervical heat treatment is a relatively new form of treatment19 where a smaller, defined area of the cervix is destroyed by insertion of a heated probe. Cervical heat treatment is already used in specialist medical practice for patients with erythroplakia, contact bleeding, chronic cervicitis and discharged. In a collaboration between Zealand and the Capital Region, 120 women are randomized to receive thermal ablation for HPV infections without severe disease with a matched control group of 120 women who do not receive ablation. All women are monitored through repeated cervical cytology re-tests at defined follow up (FU) times. The study cohort consist of 1) sample on enrollment date, 2) 3 months FU sample, 3) 6 months FU sample, 4) 12 months FU sample. All samples are collected in SurePath liquid-based cytology medium and HPV tested using the BD Onclarity HPV test (BD Integrated Diagnostic systems, Sparks, MD)20-22 supplemented by a full genotyping analysis (Seegene, Seul, Korea)21,23. Methylation status is examined using the QiaSure FAM19A4/miRNA 122-4 methylation test (Qiagen, Hilden, Germany).

This project element aims to determine whether thermal ablation impact viral clearance compared to the control group, and whether DNA methylation status is significant amongst women who are persistently HPV positive before and after thermal ablation.

ELIGIBILITY:
Inclusion Criteria:

* Women, age ≥40 years;
* persistent high-risk human papillomavirus (HR-HPV) infection for ≥12 months
* colposcopy referral according to national screening guidelines;
* normal, ASC-US, or LSIL cytology;
* no histologically verified ≥CIN2; and no prior cervical treatment.

Exclusion Criteria:

* Women with histologically confirmed ≥CIN2
* biopsies lacking transformation zone tissue

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
HPV test result after 3 and 10 months | up to 10 months follow-up post intervention
  HPV test of women after intervention or no treatment at 3 and 10 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Bonde, PhD, Study Chair — AHH-Hvidovre Hospital; Charlotte Floridon, MD, Principal Investigator — Gynecological Clinic, Holbæk
Locations (1):
- Dept. Pathology, AHH-Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared upon specific requests to the study chair. If request is compliant with current Danish Data Regulations, access will be given in form of an anonymized data sheet with all primary registered data